CLINICAL TRIAL: NCT03852979
Title: Neo-Adjuvant Chemotherapy and Conservative Surgery in Cervical Cancer to Preserve Fertility
Acronym: NEOCON-F
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study is merged with CONTESSA study
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M17CPF
Record Dates: First submitted 2017-12-05; First posted 2019-02-25 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2018-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Carboplatin; Conization

STUDY DESIGN:
Intervention Model Description: One arm two-stage Simon's design with response to neo-adjuvant chemotherapy as the primary endpoint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neo-adjuvant chemotherapy (Experimental): The patients are given weekly paclitaxel 80 mg/m2 + carboplatin AUC=2 (or AUC=6 per three weeks) during 12 weeks/4 courses followed by conization if tumor size is reduced to <2 cm
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Procedure: conisation

INTERVENTIONS:
Drug: Paclitaxel — weekly paclitaxel 80 mg/m2 for 12 weeks
Drug: Carboplatin — weekly carboplatin AUC=2 for 12 weeks
Procedure: conisation — if tumor is reduced to <2 cm, patients will be treated with a conisation

SUMMARY:
If no metastases are observed, patients will start a short protocol of four courses of weekly neo-adjuvant chemotherapy (12 weeks). If response to chemotherapy results in a tumor of less than 2 cm, cervical conisation will be performed.

DETAILED DESCRIPTION:
The standard treatment of stage Ib1 2-4 cm cervical cancer in women who wish to preserve fertility is an abdominal radical trachelectomy with pelvic lymph node dissection. Since the number of take home babies after completing this procedure is below 10%, there is a need for exploration of alternative treatment modalities with better chances of preserving fertility at equal risk of recurrence. Since low fertility rates after abdominal radical hysterectomy are observed due to the radical surgery performed on the uterine cervix, less radical surgery is warranted. To enable less radical surgery by cervical conisation, neo-adjuvant chemotherapy to reduce tumor size is incorporated to the multi-modal treatment scheme of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage Ib1 cervical cancer measuring ≥2 - ≤4 cm on physical examination and imaging in any direction
* Histologic type: squamous cell carcinoma (SCC), adeno cell carcinoma (ACC), adeno-squamous cell carcinoma (ASC)
* Lymph vascular space invasion allowed (LVSI)
* Age ≥18 years and ≤ 40 years
* Wish to preserve fertility
* Written and signed informed consent
* Negative serum or urine pregnancy test within 14 days prior to registration, and an effective method of contraception must be used during treatment
* MRI abdomen and pelvis, chest X-ray must be performed and negative for metastatic disease within 12 weeks of enrolment
* No metastases on pelvic lymph node dissection
* Laboratory values: serum creatinine < 140 μmol/L; creatinine clearance > 60 ml/min(Cockroft formula); white blood cell count > 3.5 x 109/l; platelets > 100 x 109 /l

Exclusion Criteria:

* Other high grade histologies like neuro-endocrine and clearcell carcinoma
* FIGO stage Ia, Ib1< 2 cm, Ib2, II, III and IV disease
* Involvement of tumor in uterine corpus on MRI or hysteroscopy if performed
* Evidence of metastatic disease on imagining (PET/CT/MRI) performed within 12 weeks of enrolment
* other malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
efficacy of neo-adjuvant chemotherapy | week 6 of neoadjuvant treatment
  efficacy of neo-adjuvant chemotherapy on tumor response
safety of neo-adjuvant chemotherapy | 2 years after conisation
  defined as number of women who get recurrence within two years after conisation

SECONDARY OUTCOMES:
fertility | 5 years after treatment
  number of patients who are still fertile after treatment
ovarian function | 2 years after conisation
  hormone levels will be measured to evaluate ovarian function

CONTACTS AND LOCATIONS:
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to be determined